CLINICAL TRIAL: NCT04742153
Title: A Multicenter, Non-randomized, Open-label Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG002 in the Treatment of Patients With HER2-low Locally Advanced or Metastatic Breast Cancer (BC)
Brief Title: A Study of MRG002 in the Treatment of Patients With HER2-low Locally Advanced or Metastatic Breast Cancer (BC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-005
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Advanced or Metastatic Breast Cancer
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Breast Cancer (BC)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002 (Experimental): MRG002 will be administrated via intravenous infusion of 2.6 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 in patients with HER2-low locally advanced or metastatic BC.

DETAILED DESCRIPTION:
The study will be conducted in two parts. The first part is efficacy exploration and the second part is efficacy verification. During the course of efficacy exploration, 33 subjects will be enrolled to preliminarily evaluate the safety and efficacy of MRG002. The second part will be adjusted according to the result of the first part. 29 subjects are planned to be enrolled. Considering the dropout rate of 10%, approximately 33 subjects are planned to be enrolled. A total of 66 subjects are planned to be enrolled in efficacy exploration and verification.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary to sign the ICF and follow the requirements specified in the protocol;
2. Aged ≥ 18, both genders;
3. Expected survival time ≥ 12 weeks;
4. The score of ECOG for performance status is 0 or 1;
5. Subjects with histologically confirmed HER2-low breast cancer, are currently in the locally advanced or metastatic stage, and are ineligible for radical excision, and have received at least first-line standard treatment for recurrent or metastatic breast cancer;
6. Archival or biopsy tumor specimens should be provided;
7. Subjects must have imaging evidence of tumor progression during or after the most recent treatment confirmed by the investigator and at least one measurable lesion at the baseline according to the Response Evaluation Criteria In Solid Tumors (RECIST 1.1);
8. Prior anti-tumor treatment-related AEs (NCI CTCAE v5.0 Criteria) have recovered to ≤ Grade 1 (except for alopecia, non-clinically significant or asymptomatic laboratory abnormalities);
9. No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%;
10. The level of organ functions must meet the basic requirements;
11. Reproductive male subjects and female subjects of childbearing age shall be willing to take effective contraceptive measures from the date signing the ICF to 6 months after the last dose of the IP.

Exclusion Criteria:

1. With previous history of other primary malignancies;
2. Received chemotherapy, radiotherapy, biotherapy, immunotherapy, or other anti-tumor drugs within 4 weeks prior to the first dose;
3. The subjects have central nervous system (CNS) metastasis;
4. Subjects with clinical symptoms of pleural effusion, seroperitoneum or pericardial effusion, for which treatment by puncture and drainage is required;
5. Subjects with peripheral neuropathy of greater than Grade 2 (NCI CTCAE v5.0);
6. Any severe or uncontrolled systemic disease;
7. Patients with poorly controlled heart disease;
8. Evidence of active infection, including but not limited to hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection, uncontrolled active bacterial infection, infection caused by other viruses, fungi, rickettsia or parasites;
9. History of hypersensitivity to any component of MRG002 or history of hypersensitivity of ≥ Grade 3 to trastuzumab injection;
10. Disease progression or recurrence occurred during or after the previous treatment, without evidence of CT/MRI examination results;
11. Subjects with uncontrolled concurrent diseases may have limited ability to obey the study requirements or impaired ability to sign the written ICF;
12. Subjects with active autoimmune disease or a history of autoimmune disease are receiving immunosuppressive agents or systemic hormone therapy, and are still receiving within 2 weeks prior to enrollment;
13. Received anti-tumor vaccine treatment 4 weeks prior to the first dose, or plan to participate in anti-tumor vaccine studies;
14. History of interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc;
15. Pulmonary embolism or deep vein thrombosis occurred within 3 months prior to the first dose;
16. Female subjects with positive result in serum pregnancy test, or female subjects within lactation period and do not agree to take adequate contraceptive measures during the trial and 6 months after receiving the IP;
17. Other conditions inappropriate for participation in this study, as deemed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee(IRC) | Baseline to study completion (12 months)
  ORR was defined as the proportions of subjects with a complete response (CR) and partial response (PR). ORR will be assessed by Independent Review Committee (IRC) according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Investigator | Baseline to study completion (12 months)
  ORR was defined as the proportions of subjects with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.
Progression Free Survival (PFS) | Baseline to study completion (12 months)
  PFS was defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
6-month and 12-month Progression Free Survival Rate (PFSR) | Baseline to study completion (12 months)
  The proportions of subjects surviving without progression from the start of treatment to 6-month and 12-month duration.
Time to Response (TTR) | Baseline to study completion (12 months)
  TTR was defined as the duration from the start of treatment to the first onset of CR or PR in tumor evaluation.
Duration of Response (DoR) | Baseline to study completion (12 months)
  DOR was defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Disease Control Rate (DCR) | Baseline to study completion (12 months)
  DCR was defined as the proportions of subjects achieving CR, PR, and stable disease (SD) after treatment.
Overall Survival (OS) | Baseline to study completion (12 months)
  OS was defined as the duration from the start of treatment to death of any cause.
Incidence of Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Incidence of AEs and serious adverse events (SAEs) will be assessed based on NCI-CTCAE v5.0.
Pharmacokinetics (PK) parameter for MRG002: concentration-time curve | Baseline to 14 days after decision to discontinue treatment
  Concentration-time curve will be depicted based on pharmacokinetics concentration set (PKCS).
Immunogenicity | Baseline to 14 days after decision to discontinue treatment
  The incidence of anti-drug antibody (ADA) analysis will be summarized for all patients who received at least one cycle study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, Doctor, Principal Investigator — Fifth Medical Center of PLA General Hospital; Cuizhi Geng, Doctor, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (2):
- China (2):
  - Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - The Fourth hospital of Hebei Medical University, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No